CLINICAL TRIAL: NCT03475511
Title: The Usage of High-resolution Magnetic Resonance Imaging in Patients With Disorders of Consciousness for Early Diagnosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: High-resolution MRI
Record Dates: First submitted 2018-03-18; First posted 2018-03-23 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2017-11

CONDITIONS: High-resolution Magnetic Resonance Imaging; Disorders of Consciousness
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, high-resolution brain functional magnetic resonance imaging (MRI) was used to evaluate the differences in brain structure and brain function network between patients with different degrees of disturbance of cognition and healthy controls by means of cohort follow-up and control study. The changes of patients' The dynamic changes of learning, to explore its clinical value as an early diagnosis. Combined with neurobehavioral scales and high-resolution brain structure, functional magnetic resonance imaging data to assess the brain structure, functional characteristics and consciousness of patients with impaired consciousness, and initially establish awareness of patients with recovery of consciousness Predictable imaging signs. Twenty eligible controls, 20 VS patients, and 20 MCS patients will be considered for inclusion in the inclusion / exclusion criteria. Informed consent will be obtained as required before starting any registration process.

ELIGIBILITY:
Inclusion Criteria:

(1) no use of centrally acting drugs, (2) no use of neuromuscular function blockers and no sedation within the prior 24 h, (3) periods of eye opening indicating a preserved sleep-wake cycle, and (4) a diagnosis of VS or MCS established according to internationally established criteria

Exclusion Criteria:

Magnetic resonance contraindications

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: These patients were admitted to the Department of Rehabilitation at Hangzhou Hospital of Zhejiang CAPR.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-10-15 (Actual); Primary Completion 2019-06-15 (Estimated); Study Completion 2020-01-15 (Estimated)

PRIMARY OUTCOMES:
Diffusion magnetic resonance imaging analysis | Three months
  The color-coding of tractography pathways in was determined for a visualization purpose. The color-coding of tractography pathways was based on FA values.

CONTACTS AND LOCATIONS:
Overall Officials: Benyan F Luo, MD, Principal Investigator — Department of Neurology and Brain Medical Centre The First Affiliated Hospital, School of Medicine, Zhejiang University 79 Qingchun Road, Hangzhou; Jian M Gao, Principal Investigator — Hangzhou Hospital of Zhejiang CAPR,Hangzhou, Zhejiang, China
Locations (1):
- Hangzhou Hospital of Zhejiang CAPR, Hangzhou, Zhejiang, China